CLINICAL TRIAL: NCT01553422
Title: Assessment of Relation Between Intrabdominal Pressure and Collapsibility Index of Inferior Vena Cava by Emergency Ultrasonography Before and After Fluid Therapy
Brief Title: Relation Between Intrabdominal Pressure and Collapsibility Index of Inferior Vena Cava Before and After Fluid Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Keihan Golshani, Assistant Professor of Emergency Medicine, Director of Emergency Medicine Residency Program, Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 390331
Record Dates: First submitted 2012-03-07; First posted 2012-03-14 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Abdominal Compartment Syndrome
Keywords: Intrabdominal Pressure; Emergency Bedside Ultrasonography; Abdominal Compartment Syndrome
MeSH Terms: conditions — Intra-Abdominal Hypertension | interventions — Fluid Therapy; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- before fluid Therapy (Active Comparator)
  Interventions: Other: Fluid therapy (Saline Normal)
- after fluid Therapy (Active Comparator)
  Interventions: Other: Fluid therapy (Saline Normal)

INTERVENTIONS:
Other: Fluid therapy (Saline Normal) — Saline Normal 1 Lit. during 30 minutes
  Arms: before fluid Therapy
Other: Fluid therapy (Saline Normal) — saline Normal 1 lit during 30 minutes
  Arms: after fluid Therapy

SUMMARY:
This study assess the relation between intra abdominal pressure and collapsibility index of inferior vena cava in emergency bedside ultrasonography before and after fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index less than 30
* Written agree of the patient to participate in the study

Exclusion Criteria:

* neurogenic bladder or any documented previous surgery on bladder, spastic or contractile bladder
* large abdominal hernia
* patients who received neuromuscular blocking agents
* Patients with abdominal respiration due to chest pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Emergency bedside Ultrasonography assessment of Inferior Vena cava collapsibility index before and after fluid therapy | "up to 36 weeks"

CONTACTS AND LOCATIONS:
Overall Officials: KEIHAN GOLSHANI, M.D., Study Chair — Isfahan University of Medical Sciences
Locations (1):
- Emergency department, Alzahra General Hospital, Isfahan, Isfahan, Iran